CLINICAL TRIAL: NCT04617457
Title: Open-label, Single Arm Phase II Trial Investigating the Efficacy, Safety and Quality of Life of Neoadjuvant Chemotherapy With Liposomal Irinotecan Combined With Oxaliplatin and 5-Fluorouracil/Folinic Acid Followed by Curative Surgical Resection in Patients With Hepatic Oligometastatic Adenocarcinoma of the Pancreas
Brief Title: Chemotherapy and Surgical Resection in Patients With Hepatic Oligometastatic Adenocarcinoma of the Pancreas
Acronym: HOLIPANC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Collaborators: Servier (Industry)
Responsible Party: Principal Investigator, Florian Gebauer, Principal investigator, University of Witten/Herdecke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-4067; 2019-002734-37 (EudraCT Number); 20-1544-AMG (Other: Local Ethics Committee University of Cologne)
Record Dates: First submitted 2020-10-29; First posted 2020-11-05 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Pancreatic Cancer; Metastasis; Surgery; Oligometastatic Disease
Keywords: pancreatic cancer; NAPOX; chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — irinotecan sucrosofate; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NAPOX chemotherapy (Experimental): NAPOX chemotherapy in 14-day cycles with the four IMPs given intravenously in the following order: nal-irinotecan, oxaliplatin, folinic acid and 5-fluouracil.
  Interventions: Drug: nal-irinotecan (nal-iri) (Onyvide), oxaliplatin (ox), 5-fluouracil (5-FU), folinic acid (FA)

INTERVENTIONS:
Drug: nal-irinotecan (nal-iri) (Onyvide), oxaliplatin (ox), 5-fluouracil (5-FU), folinic acid (FA) — preoperative chemotherapy
  Other Names: nal-irinotecan (nal-iri); oxaliplatin (ox); 5-fluouracil (5-FU); folinic acid (FA); ONIVYDE TM

SUMMARY:
This is an interventional, open-label, non-randomised, multicentre, single-arm phase II clinical trial.

Eligible patients with hepatic oligometastatic adenocarcinoma of the pancreas will receive neoadjuvant combination chemotherapy (liposomal irinotecan, oxaliplatin, 5-fluouracil, folinic acid (NAPOX)) in cycles of 14 days. Patients with tumour response or stable disease and a resectable primary tumour after the first 4 cycles will undergo explorative laparotomy and synchronous resection of the tumour and hepatic metastases, if feasible; these patients may receive 4 more cycles of neoadjuvant chemotherapy 2-4 weeks after the explorative laparotomy if the surgeon rated the primary tumour as non-resectable during the explorative laparotomy.

DETAILED DESCRIPTION:
This is an interventional, open-label, non-randomised, multicentre, single-arm phase II clinical trial.

Eligible patients with hepatic oligometastatic adenocarcinoma of the pancreas will receive neoadjuvant NAPOX chemotherapy in cycles of 14 days.

In patients with progressive disease during or after the first 4 cycles, neoadjuvant chemotherapy will be permanently discontinued. Patients with tumour response or stable disease after the first 4 cycles according to RECIST v1.1 but a non-resectable primary tumour according to the evaluation of an interdisciplinary tumour board will receive 4 more cycles of neoadjuvant chemotherapy. Patients with tumour response or stable disease and a resectable primary tumour after the first 4 cycles will undergo explorative laparotomy and synchronous resection of the tumour and hepatic metastases, if feasible; these patients may receive 4 more cycles of neoadjuvant chemotherapy 2-4 weeks after the explorative laparotomy if the surgeon rated the primary tumour as non-resectable during the explorative laparotomy.

All patients who receive a total of 8 cycles and who then have tumour response or stable disease according to RECIST v1.1 will undergo exploratory laparotomy surgery and synchronous resection of the tumour and hepatic metastases, if feasible according to the surgeon, 2-6 weeks after the last investigational medicinal product (IMP) treatment.

The primary endpoint of the clinical trial is overall survival of patients with an R0/R1 resection after neoadjuvant chemotherapy.

The IMP treatment will be discontinued if tumour progression or inacceptable toxicity occurs or other termination criteria apply.

Adjuvant treatment will not be part of the trial treatment and may be given at the investigator's discretion in accordance with the Onkopedia guideline for pancreatic cancer.

Tumour, stool and blood samples will be collected before start and during the clinical trial for translational research if the patient gives his/her consent to participating in the translational research programme.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of treatment-naïve limited hepatic metastatic adenocarcinoma of the pancreas Definition of limited hepatic metastasis: 1 to 5 metastases in CT/MRI and/or contrast-enhanced ultrasound scan, which are potentially resectable or treatable by ablative procedures (Note 1: Patients also fulfil this inclusion criterion if a hepatic metastasis was partly or entirely removed as part of the diagnosis and is thus not detectable by CT/MRI and/or contrast-enhanced ultrasound scan at screening. Note 2: If more than 5 metastases are unexpectedly detected during surgery, it is not a violation of this inclusion criterion if the excess metastases had not been detectable by CT/MRI and/or contrast-enhanced ultrasound scan at screening.)
2. Measurable disease according to RECIST v1.1
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
4. Adequate renal, hepatic and bone marrow function, defined as

   * Calculated creatinine clearance ≥60 mL/min
   * Total bilirubin ≤2 mg/dL; patients with biliary stent may be included if bilirubin level decreased to ≤2 mg/dL after stent insertion
   * alanin-aminotransferase and aspartat-aminotransferase (ALT and AST) ≤5 × upper limit of normal (ULN)
   * Absolute neutrophil count (ANC) ≥1.5 × 109/L
   * Thrombocytes ≥100 × 109/L
   * Haemoglobin ≥9 g/dL
   * activated partial thromboplastin time (aPTT) ≤1.5 × ULN and Quick value ≥70%
5. Patients ≥18 years at the time of signing the informed consent
6. Females of childbearing potential (FCBPs) must agree to use highly effective contraceptive measures (Pearl index <1) or practice true abstinence from any heterosexual intercourse for the duration of treatment and for at least 1 month after the last IMP administration (true abstinence is acceptable when this is in line with the preferred and usual lifestyle of the patient). A woman will be considered as being of childbearing potential unless she is at least 50 years old and, moreover, has gone through menopause for at least 2 years or has been surgically sterilised.
7. Males must agree to use condoms or practice true abstinence from any heterosexual intercourse for the duration of IMP treatment and at least 6 months after the last IMP administration (true abstinence is acceptable if this is in line with the patient's preferred and usual lifestyle). Male patients must furthermore refrain from donating sperm during the clinical trial until at least 6 months after the last IMP administration.
8. Patient's written informed consent prior to any trial-specific procedure
9. Patient's legal capacity to consent to participation in the clinical trial

Exclusion Criteria:

1. Acinar cell carcinoma and/or neuroendocrine carcinoma of the pancreas
2. Symptomatic clinically significant ascites
3. Evidence of any distant metastases other than limited hepatic metastasis as defined in inclusion criterion 1
4. Any tumour-specific pretreatment of the adenocarcinoma of the pancreas (including but not limited to surgery, radiation therapy, chemotherapy or ablative procedures)
5. Any malignancies other than adenocarcinoma of the pancreas in the 5 years before the start of the clinical trial except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, breast cancer, prostate cancer or superficial bladder tumours (Ta, Tis and T1)
6. Hypersensitivity to any of the IMPs or any of the excipients
7. Any major surgery within 4 weeks before the first IMP administration
8. Pregnant or breast-feeding female
9. Known chronic inflammatory bowel disease, bowel obstruction or chronic diarrhoea Grade ≥2 according to NCI CTCAE version 5.0
10. Peripheral polyneuropathy Grade ≥2 according to NCI CTCAE version 5.0
11. Known interstitial lung disease (ILD) or pulmonary fibrosis
12. Radiographic evidence of severe portal hypertension
13. Liver cirrhosis ≥ Child Pugh B
14. Cholestasis or cholangitis despite adequate biliary stenting; treatment with anti-infectious agents is permitted; patient must be disease-free and without anti-infectious treatment for 7 days before the first IMP administration
15. Active infection requiring systemic therapy
16. Known HIV seropositivity
17. Active or chronic Hepatitis B or Hepatitis C infection
18. Known glucuronidation deficiency (Gilbert's syndrome) (specific screening not required)
19. Known complete dihydropyrimidine dehydrogenase (DPD) deficiency (specific screening according to the recommendations of the Summary of Product Characteristics (SmPC) in effect for 5-FU; patients with a known complete DPD deficiency must be excluded; patients with a known partial DPD deficiency may be included
20. Clinically significant cardiovascular or vascular disease or disorder ≤6 months before enrolment into the clinical trial (e.g. myocardial infarction, unstable angina pectoris, chronic heart failure New York Heart Association (NYHA) ≥ Grade 2, uncontrolled arrhythmia, cerebral infarction)
21. Pulmonary embolism, deep venous thrombosis or arterial thromboembolism ≤6 months before before the first IMP administration
22. Any other severe concomitant disease or disorder, which could influence patient's ability to participate in the clinical trial and his/her safety during the trial or interfere with interpretation of results; e.g., severe hepatic, renal, pulmonary, cardiovascular, metabolic or psychiatric disorders
23. Requirement for live vaccination within 4 weeks before the first IMP administration and during neoadjuvant chemotherapy
24. Use of strong CYP3A4 inhibitors (Strong CYP3A4 inhibitors have to be discontinued at least one week prior to start of trial treatment.); use of strong UGT1A1 inhibitors or strong CYP3A4 inducers unless there are no therapeutic alternatives
25. Treatment with nucleoside analogues such as brivudine within 4 weeks before the first IMP administration or requirement for concomitant antiviral treatment with brivudine or analogues
26. Participation in a clinical trial or experimental drug treatment within 4 weeks before the first IMP administration or within a period of 5 half-lives of the substances administered in a clinical trial or during an experimental drug treatment before the first IMP administration, depending on which period is longest, or simultaneous participation in another clinical trial while taking part in this clinical trial
27. Continuing abuse of alcohol, drugs or medical drugs
28. Patient committed to an institution by virtue of an order issued either by the judicial or the administrative authorities
29. Patients possibly dependent from the investigator including the spouse, children and close relatives of any investigator at the discretion of the investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival after R0/R1 resection (OS-res) | max 24 months follow-up
  OS for patient after macroscopic tumor resection

SECONDARY OUTCOMES:
R0/R1 resection rate after neoadjuvant chemotherapy | direct after operation
  Fraction of patients that undergo macroscopically complete tumor resection (No and %)
Overall survival (OS) | max 24 months follow-up
  time from study inclusion until death (months)
Progression-free survival (PFS) after R0/R1 resection according to RECIST v1.1 | max 24 months follow-up
  time from study inclusion until tumor progress/recurrence (months)
Type, frequency and severity of adverse events (AE) with severity (SAE) according to NCI CTCAE version 5.0 | direct after IMP administration up to 3 months after completion of study
  Number and fraction of AE/SAEs (No and %)
HR-QoL according to EORTC QLQ-C30 | 90 days after operation
  Quality of Life according to the EORTC QLQ-C30 questionaire (scale 0 (poor) - 7 (excellent)
Quality of life (QoL) according to EORTC QLQ-PAN-26 | 90 days after operation
  Quality of Life according to the EORTC QLQ-PAN26 questionaire (scale 0 (poor) - 7 (excellent)
QoL-adjusted OS | max 24 months follow-up
  time from study inclusion until death (months) adjusted to quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Florian Gebauer, MD, Principal Investigator — University of Witten/Herdecke; Dirk Waldschmidt, Study Director — University of Cologne
Locations (11):
- Germany (11):
  - University Aachen, Aachen
  - University of Berlin, Charité, Campus Benjamin-Franklin, Berlin
  - University of Bonn, Bonn
  - Städtisches Klinikum Dresden, Dresden
  - University of Düsseldorf, Düsseldorf
  - University of Freiburg, Freiburg im Breisgau
  - University of Halle (Saale), Halle
  - University of Heidelberg, Heidelberg
  - Klinikum Großhadern, LMU München, München
  - Klinikum Rechts der Isar Technische Universität München, München
  - University of Regensburg, Regensburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gebauer F, Damanakis AI, Popp F, Quaas A, Kutting F, Lutz K, Held S, Deuss B, Goser T, Waldschmidt D, Bruns C. Study protocol of an open-label, single arm phase II trial investigating the efficacy, safety and quality of life of neoadjuvant chemotherapy with liposomal irinotecan combined with Oxaliplatin and 5-fluorouracil/Folinic acid followed by curative surgical resection in patients with hepatic Oligometastatic adenocarcinoma of the pancreas (HOLIPANC). BMC Cancer. 2021 Nov 18;21(1):1239. doi: 10.1186/s12885-021-08966-3. PMID 34794396